CLINICAL TRIAL: NCT01946815
Title: Phase 3 Study of Effect of ATorvastatin on Fractional Flow Reserve in Coronary Artery Disease
Brief Title: Effect of Atorvastatin on Fractional Flow Reserve in Coronary Artery Disease
Acronym: FORTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Ulsan University Hospital (Other); Inje University Ilsan Paik Hospital (Other)
Responsible Party: Principal Investigator, NAM, Chang-Wook, Associate Professor of Internal Medicine, Keimyung University Dongsan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FORTE
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin (Experimental): Atorvastatin (Lipitor) will be prescribed with 20mg,40mg,or 80mg by the unit of 28 tablets upon the result of lipid profile. Besides Clinical and lab test, follow-up CAG, IVUS(optional) and FFR will be performed in 12 months.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Lipitor dose titration will be followed by the result of LDL lab test until it meets the target level of LDL. IVUS(optional) and FFR during follow up CAG in 12 months will be measured to evaluate the effect of lipitor.
  Other Names: lipitor

SUMMARY:
Natural course of intermediate coronary artery disease (CAD) is very important to predict the prognosis of the patient with such disease.

Several studies have well demonstrated the beneficial effect of lipid-lowering therapy on the progression of CAD with the modification of lipid profiles.

This effect can be also explained by intravascular ultrasound (IVUS) or optical coherence tomography. However, the effect of plaque modification on coronary physiology has been rarely evaluated.

This research is to evaluate the change of intermediate or nonculprit coronary lesion on lipid-lowering therapy via IVUS(optional) and FFR.

DETAILED DESCRIPTION:
The patients who have intermediate CAD (30-80% diameter stenosis by visual estimation) with FFR≥0.80, or nonculprit coronary artery disease with FFR≥0.8 after culprit coronary artery disease intervention will be enrolled. FFR, IVUS(optional) and index of microcirculatory resistance (IMR) should be performed simultaneously. Atorvastatin 20mg is a starting dose, then up-titration will be done twice within each 4~6weeks until LDL target goal (① LDL<70mg/dl, or ② statin naive: >50% reduction from baseline LDL, current statin user: >30% reduction from baseline LDL). First titration will be atorvastatin 40mg, second will be atorvastatin 80mg. If patients have any adverse effect on atorvastatin, the dose of atorvastatin can be adjusted by investigator's decision. Official clinical follow-up except visit for statin dose titration will occur at 1, 12 months after index procedure. Follow-up coronary angiography, FFR,IMR,and IVUS(optional) will be performed 12 months after index procedure.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years of age and willing to participate
* patients who have stable intermediate CAD(30-80% diameter stenosis by visual estimation) on angiography with FFR≥0.8,or who have nonculprit CAD which is not planned revascularization
* Signed written Informed Consent

Exclusion Criteria:

* Patients who are in cardiogenic shock
* Patients with LVEF<35%
* Patients with left main disease, restenotic, bypass grafted lesions
* Patients with platelet count < 100,000 cell/mm3
* Patients who have co-morbidity which reduces life expectancy to one year
* Patients who have a history of stroke or transient ischemic attack within 6 months
* Patients who are planned discontinuation of medication due to surgery
* Patients with known adverse reaction to HMG CO-A reductase therapy (statins)
* Patients with liver disease (elevation of AST or ALT more than 2 times)
* Patient with creatinine > 2.0 mg/dL
* Pregnant women and women of childbearing potential who intend to have children during the duration of the trial
* Patients who consistently must take drugs affecting lipid levels in blood except the investigational product

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-09; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
changes of FFR between baseline and 12months follow-up | up to 1 year
  changes of FFR(fractional flow reserve) baseline and 12month foloow-up

SECONDARY OUTCOMES:
Change of FFR according to the degree of decreased LDL | up to 1 year
  Change of FFR according to the degree of decreased LDL
Change of % plaque volume, total atheroma volume & plaque compositions in lesion of interest | up to 1 year
  Change of % plaque volume, total atheroma volume & plaque compositions in lesion of interest
Change of IMR | up to 1 year
  Change of IMR(index of microcirculatory resistance)
Death including cardiac and noncardiac | up to 1 year
  Death including cardiac and noncardiac
Myocardial infarction | up to 1 year
  Myocardial infarction
Target lesion and vessel revascularization rate | up to 1 year
  Target lesion and vessel revascularization rate
CVA: hemorrhage and infarction | up to 1 year
  CVA(cerebrovascular accident): hemorrhage and infarction
side effect of statin : liver and muscle enzyme | up to 1 year
  side effect of statin : liver and muscle enzyme

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Wook Nam, Postdoctoral, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (4):
- South Korea (4):
  - Ulsan University Hospital, Ulsan, Gyeongsangbuk-do
  - Inje University Ilsan Paik Hospital, Ilsan, Kyeongki
  - Keimyung University Dongsan Medical center, Daegu
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Lee CH, Hwang J, Kim IC, Cho YK, Park HS, Yoon HJ, Kim H, Han S, Hur SH, Kim KB, Kim JY, Chung JW, Lee JM, Doh JH, Shin ES, Koo BK, Nam CW. Effect of Atorvastatin on Serial Changes in Coronary Physiology and Plaque Parameters. JACC Asia. 2022 Nov 1;2(6):691-703. doi: 10.1016/j.jacasi.2022.07.010. eCollection 2022 Nov. PMID 36444331